CLINICAL TRIAL: NCT05541250
Title: Safety and Efficacy of Autologous Human Schwann Cell (ahSC) Augmentation in Severe Peripheral Nerve Injury (PNI)
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: W. Dalton Dietrich (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency)
Responsible Party: Sponsor-Investigator, W. Dalton Dietrich, Professor, University of Miami
Organization: University of Miami (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 20220447; OR210075 (Other Grant/Funding Number: United States Department of Defense)
Record Dates: First submitted 2022-09-13; First posted 2022-09-15 (Actual); Last update posted 2025-09-02 (Actual); Status verified 2025-08

CONDITIONS: Peripheral Nerve Injury
MeSH Terms: conditions — Peripheral Nerve Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Autologous Human Schwann Cell (ahSC) Group (Experimental): Participants in this group will undergo a sural nerve biopsy followed by ahSC transplant
  Interventions: Biological: Autologous Human Schwann Cell

INTERVENTIONS:
Biological: Autologous Human Schwann Cell — A one-time dose of 1000 μl* or 80 to 100 million ahSC prepared from segments of the sural nerve from the leg recovered from the participant.

SUMMARY:
The primary purpose of this research study is to evaluate the safety and possible harms of injecting one's own Schwann cells along with nerve auto-graft after a severe injury to a major nerve has occurred.

ELIGIBILITY:
Inclusion Criteria:

1. Persons with severe sciatic nerve injury, brachial plexus injury, and/or major nerve injury at the upper or lower extremity within previous year;
2. Between the ages of 18 and 65 at last birthday

Exclusion Criteria:

1. Persons unable to safely undergo an MRI;
2. Persons with pre-existing conditions that would preclude satisfactory sural nerve harvest;
3. Persons with severe peripheral nerve injury gap length > 10 cm;
4. Persons with history of radiation or local cancer in area of nerve injury, including primary tumors of the nerve;
5. Pregnant women or a positive pregnancy test in those women with reproductive potential prior to enrollment;
6. Presence of disease that might interfere with participant safety, compliance, or evaluation of the condition under study;
7. History of active substance abuse;
8. Persons allergic to gentamicin;
9. Persons who test positive for HIV or Hepatitis B or C virus.
10. Persons unable to provide consent independently due to cognitive impairment

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-05-04 (Actual); Primary Completion 2026-09-29 (Estimated); Study Completion 2026-09-29 (Estimated)

PRIMARY OUTCOMES:
Incidence of Treatment-related Adverse Events (AEs) | Up to 2 years
  Safety will be reported as the incidence of treatment-related AEs as assessed by treating physician

SECONDARY OUTCOMES:
Motor Recovery as assessed using the MRC Grading Scale | Up to 2 years
  Motor recovery will be assessed using the Medical Research Council (MRC) Grading Scales. MRC Grading Scale scores ranges from 0-5 with a higher score indicating better function
Sensory recovery as assessed by Pin-Prick Evaluation | Up to 2 years
  Pin prick evaluation will be assessed using the Semmes Weinstein Monofilament Evaluation. Semmes Weinstein Monofilament evaluation has a total score ranging from 0-5 with a higher score indicating better function
Sensory recovery as assessed by the 2-Point Discrimination Evaluation | Up to 2 years
  2-Point Discrimination Evaluation scoring ranges from 2-20mm with a higher score indicating worse function

CONTACTS AND LOCATIONS:
Overall Officials: W. Dalton Dietrich, MD, Study Chair — University of Miami
Locations (1):
- University of Miami, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No